

## **MP17 Statistical Analysis Plan**

Version 1: 14 February 2018

Version 2: 03 September 2019

SPONSOR Multidisciplinary Association for Psychedelic Studies (MAPS)

1115 Mission Street Santa Cruz, CA 95060

SPONSOR Rick Doblin, Ph.D.

REPRESENTATIVE Executive Director, MAPS

SPONSOR DELEGATE &

TRIAL ORGANIZER

MAPS Public Benefit Corporation (MPBC)

1115 Mission Street

Santa Cruz, CA 95060

SPONSOR DESIGNEE Amy Emerson

Executive Director and Director of Clinical Research, MPBC

Phone number: 510-393-7224 Email: <a href="mailto:amy@mapsbcorp.com">amy@mapsbcorp.com</a>

MEDICAL MONITOR(S)

STATISTICIAN(S)

Michael Mithoefer, M.D. Scott Hamilton, Ph.D.

PREPARED BY Scott Hamilton, Ph.D.

Allison Feduccia, Ph.D. Berra Yazar-Klosinski, Ph.D.

Ilsa Jerome, Ph.D.

USE In conjunction with relevant FDA and HC guidance

# **Table of Contents**

| List of Tables | 3 |
|-------------------------------------------------------|----|
| List of Abbreviations | 4 |
| 1.0 Definitions of Terms | 7 |
| 2.0 Introduction | |
| 3.0 Study Objectives | 8 |
| <b>3.1</b> Primary Objective | 8 |
| <b>3.2</b> Secondary Objective | 8 |
| <b>3.3</b> Safety Objectives | 8 |
| <b>3.4</b> Exploratory Objectives | 9 |
| 4.0 Measures | 10 |
| <b>4.1</b> Primary Measure | 10 |
| <b>4.2</b> Secondary Outcome Measure | 10 |
| <b>4.3</b> Safety Measures | |
| <b>4.4</b> Exploratory Measures | 10 |
| 5.0 Study Design | 10 |
| 6.0 Randomization and Blinding | 15 |
| 7.0 Sample Size and Power Considerations | |
| 8.0 Analyses | 15 |
| <b>8.1</b> Analysis Sets | |
| 8.2 Missing Data Handling | 15 |
| 8.2.1 Partial or Missing Dates | |
| <b>8.3</b> Protocol Deviations | |
| 8.4 Baseline Values | |
| <b>8.5</b> Participant Disposition and Dosing Summary | 17 |
| <b>8.6</b> Demographics and Baseline Characteristics. | |
| <b>8.7</b> Effectiveness Analyses | |
| 8.7.1 Primary Effectiveness Analyses | |
| 8.7.2 Key Secondary Effectiveness Analyses | 19 |
| 8.7.3 Exploratory Analyses | |
| 8.7.4 Responder Analyses | |
| 8.8 Safety Analyses | 22 |
| 8.8.1 Analysis of Exposure | 22 |
| 8.8.2 Analysis of Adverse Events | 22 |
| 8.8.3 Concomitant Medications | |
| 8.8.4 Analysis of Suicidal Ideation and Behavior | |
| 8.8.5 Summary of Vital Signs. | |
| 9.0 Timing of Analyses | 23 |

# **List of Tables**

| Table 1: Dose Regimen of MDMA | 10 |
|---------------------------------------------|----|
| Table 2: Time and Events – Study Procedures | 12 |
| Table 3: Time and Events – Study Measures | |

#### List of Abbreviations

° C Degrees Celsius A:G Albumin:Globulin

ACE Adverse Childhood Experiences Questionnaire
ADHD Attention Deficit/Hyperactivity Disorder

AE Adverse Event

AED Automatic External Defibrillator AESI Adverse Event of Special Interest

ALT Alanine Aminotransferase
AMI Acute Myocardial Infarction
API Active Pharmaceutical Ingredient
AST Aspartate Aminotransferase

AUDIT Alcohol Use Disorders Identification Test

BDI-II Beck Depression Inventory-II

BLS Basic Life Support
BMI Body Mass Index
BP Blood Pressure
BUN Blood Urea Nitrogen

CAPS-4 Clinician-Administered PTSD Scale for DSM-4 CAPS-5 Clinician-Administered PTSD Scale for DSM-5

CBC Complete Blood Count

%CDT %Carbohydrate-deficient Transferrin CMC Chemistry Manufacturing and Control

CPGS Chronic Pain Grade Scale
CRA Clinical Research Associate

C-SSRS Columbia-Suicide Severity Rating Scale
DDIS Dissociative Disorders Interview Schedule

DID Dissociative Identity Disorder

dIGPP Cohen's d Independent Groups Pre-test Post-test

DMF Drug Master File

DSM-5 Diagnostic and Statistical Manual of Mental Disorders, 5<sup>th</sup> edition

DSP-I Dissociative Subtype of PTSD Interview DUDIT Drug Abuse Disorders Identification Test

EAT-26 Eating Attitudes Test ECG Electrocardiogram

eCRF Electronic Case Report Form
ECT Electroconvulsive Therapy
ED Emergency Department
EDC Electronic Data Capture

EMDR Eye Movement Desensitization and Reprocessing

EMS Emergency Medical Services

ePRO Electronic Participant Reported Outcome

EQ-5D-5L EuroQol Five Dimensions – Five Levels Questionnaire

FDA Food and Drug Administration

GCP Good Clinical Practice

GMP Good Manufacturing Practice

HCV Hepatitis C Virus

HIV Human Immunodeficiency Virus

HIPAA Health Insurance Portability and Accountability

HPA Hypothalamic-pituitary-adrenal HPMC Hydroxypropyl Methylcellulose

HPOSF Health and Work Performance Absenteeism and Presenteeism Short Form

IASC Inventory of Altered Self-Capacities

IB Investigator's Brochure

ICD International Classification of Disease

ICF Informed Consent Form

ICH International Conference on Harmonisation

IND Investigational New Drug
IP Investigational Product

IPF Inventory of Psychosocial Functioning

IR Independent Rater

IRB Institutional Review Board
ISF Investigator Site File
ITT Intent-to-Treat
IUD Intrauterine Device

IUS Intrauterine Hormone-releasing System

kg Kilogram

LEC-5 Life Events Checklist LTFU Long-term Follow-up

MAPS Multidisciplinary Association for Psychedelic Studies

MAOI Monoamine Oxidase Inhibitor MCH Mean Corpuscular Hemoglobin

MCHC Mean Corpuscular Hemoglobin Concentration

MCV Mean Corpuscular Volume

MDMA 3,4-methylenedioxymethamphetamine MedDRA Medical Dictionary for Regulatory Activities

mg Milligram

mITT Modified Intent-to-Treat mmHg Milligrams of Mercury

MMRM Mixed Model Repeated Measure MPBC MAPS Public Benefit Corporation

ms Millisecond

PCL-5 PTSD Checklist for DSM-5

PTCA Percutaneous Transluminal Coronary Angioplasty

PTSD Posttraumatic Stress Disorder

RACT Risk Assessment and Categorization Tool

RBC Red Blood Cell

RDW Red Cell Distribution Width SAE Serious Adverse Event

SCID-5-PD Structured Clinical Interview for DSM-5 Personality Disorders

SCID-5-SPQ SCID-5 Self-report Personality Questionnaire

SCS Self-compassion Scale SDS Sheehan Disability Scale

SGOT Serum Glutamic Oxaloacetic Transaminase SNRI Serotonin-norepinephrine Reuptake Inhibitor SPGT Serum Glutamic Pyruvic Transaminase

SRNU Self-reported Nicotine Use SSR Sample size re-estimation

SSRI Selective serotonin reuptake inhibitor

SUBJID Subject Identifier

TAS-20 Toronto Alexithymia Scale

TEAE Treatment Emergent Adverse Event
TSH Thyroid-stimulating Hormone

UFEC Utilization of Facility-based and Emergent Care

U.S. United States

VA U.S. Department of Veterans Affairs

Visual Analog Scale White Blood Cell VAS WBC

WHO

World Health Organization
WHO Drug Dictionary Enhanced<sup>TM</sup> WHO DDE

#### 1.0 Definitions of Terms

Categorical data: refers to discrete (indivisible) variables, such as gender or ethnicity; data will be presented as total numbers of each category as needed to describe the sample

Completers: are defined as participants who complete all three planned experimental sessions and the CAPS-5 outcome assessment 18 weeks after randomization (Visit 19).

Descriptive data: includes mean, median, standard deviation, minimum, and maximum of numerical data used as needed to describe the sample

*Difference scores*: consist of scores computed by subtracting one value from another, as subtracting Baseline from follow-up score, used to test for differences between and within groups to determine change as a function of experimental treatment over time

*Dropouts:* are defined as participants who withdraw consent due to any reason after dosing and no longer participate in the study, i.e. no further contact with investigators or site staff.

Effectiveness: type of analysis used to assess therapeutic effects or benefits

Exploratory analyses: inferential or descriptive analysis of the data to determine trends that might lead to hypotheses for further study

Frequency listing: tabular listing of numbers and/or percentages of events used as needed to describe the sample or data characteristics

*Outcome measures*: primary and secondary study measures that are used to test the study hypotheses

*Post-dosing Early Terminators:* are defined as participants who discontinue study treatment but continue to participate in study evaluations and outcome assessments.

*Pre-dosing Early Terminators:* are defined as participants who discontinue participation after enrollment but before randomization during the Preparatory Period and never receive study drug.

*Process measures*: study measures or qualitative observations collected during the study that may increase depth of understanding of the condition and treatment, although not necessarily related to safety or effectiveness

*Protocol deviation*: event that represents significant divergence from the intended study design as described in the protocol

Safety: assessment of indicators of potential risks and adverse events

Safety measures: study measures that assess safety of the Investigational Product (IP), such as heart rate monitoring, blood pressure, body temperature

*Study design*: all elements of a research project that define the study question, experimental methods, study procedures including randomization and blinding, measurement techniques, data workflow, and statistical analysis

*Tabular listing*: list of each variable or item for each individual participant either in total or by treatment group in a table format

## 2.0 Introduction

This document contains a Statistical Analysis Plan (SAP) for MP17, "An Open-Label, Multi-Site Phase 2 Study of the Safety and Effect of Manualized MDMA-Assisted Psychotherapy for the Treatment of Severe Posttraumatic Stress Disorder."

MP17 tests a flexible dosing regimen of 100 mg MDMA in Session 1, and 100 mg or 125 mg MDMA in Sessions 2 and 3, each followed by a supplemental half-dose.

The Multidisciplinary Association for Psychedelic Studies (MAPS) is a non-profit research and educational organization working to obtain approval for the prescription use of 3,4-methylenedioxymethamphetamine (MDMA) in conjunction with psychotherapy in persons with posttraumatic stress disorder (PTSD). MAPS has delegated trial organization activities to its wholly owned subsidiary, MAPS Public Benefit Corporation (MPBC).

This open-label Phase 2 study will serve as a lead-in to the sponsor's two planned Phase 3 studies, only sites planned for Phase 3 will participate in these studies. This open-label lead-in Phase 2 study will serve to validate assumptions made for statistical power calculations supporting planned Phase 3 clinical trials and will provide data on the updated version of the instrument for the Primary Outcome measure, the Clinician Administered PTSD Scale for DSM-5 (CAPS-5), which will be used in Phase 3. In addition, this study will gather supportive data on the safety and effect of manualized MDMA-assisted psychotherapy while providing an opportunity for clinical supervision to planned Phase 3 therapy teams. This study will be the sponsor's first multi-site studies of MDMA-assisted psychotherapy for PTSD and will explore reproducibility of findings in a multi-site format to confirm the Phase 3 study design.

This version 2 of the Statistical Analysis Plan was modified from version 1. The changes made include the following, 1) separate plans were made for each individual study, MP16 and MP17; 2) analyses were modified to be within-subject and not comparison between studies; and 3) doses used in each study were updated.

#### 3.0 Study Objectives

#### 3.1 Primary Objective

The primary objective of this study is to evaluate the effect of MDMA-assisted psychotherapy on PTSD, as measured by the change in CAPS-5 Total Severity Score from Baseline (Visit 3) to 18 weeks post Baseline (Visit 19).

#### 3.2 Secondary Objective

The secondary objective is to evaluate the effect of MDMA-assisted psychotherapy for PTSD in clinician-rated functional impairment, as measured by the mean change in Sheehan Disability Scale (SDS) item scores from Visit 3 (Baseline) to Visit 19 (18 weeks post Baseline).

## 3.3 Safety Objectives

The overall safety objective is to assess severity, incidence and frequency of AEs, AEs of Special Interest (AESIs), and Serious Adverse Events (SAEs), concomitant medication use, suicidal ideation and behavior, and vital signs to support the package insert for MDMA-assisted

psychotherapy. The following safety objectives will evaluate the safety of MDMA-assisted psychotherapy.

- Assess incidence of AEs during Experimental Sessions that may be indicative of a
  medical complication of the Investigational Product (IP), such as clinical signs and
  symptoms of chest pain, shortness of breath, or neurological symptoms or any other signs
  or symptoms that prompt additional vital sign measurements.
- Assess incidence of AEs by severity.
- Assess incidence of Treatment Emergent AEs (TEAEs) by severity.
- Assess incidence of TEAEs by severity taken during an Experimental Session and 2 days after IP administration.
- Assess incidence of AESIs, defined as AEs specified in the protocol related to cardiac function and abuse liability.
- Assess incidence of AEs by severity categorized as leading to discontinuation of IP, resulting in death or hospitalization, and continuing at Termination.
- Assess incidence of SAEs.
- Assess incidence of psychiatric concomitant medications taken during an Experimental Session and 2 days after IP administration.
- Assess incidence of any psychiatric concomitant medications taken during the Treatment Period.
- Assess incidence of serious suicidal ideation and positive suicidal behavior assessed with the Columbia Suicide Severity Rating Scale (C-SSRS).
   Assess mean changes in blood pressure, heart rate, and body temperature from pre-IP administration to end of each Experimental Session.

## 3.4 Exploratory Objectives

These objectives may be used to characterize participants receiving MDMA-assisted psychotherapy to support the primary objective and to further explore the effects of treatment:

- 1. Explore the effect of presence of secondary traumatic stressors (LEC-5) on the CAPS-5 Total Severity analyses
- 2. Explore changes within-participants in PTSD symptom clusters of re-experiencing, avoidance, negative alterations in cognition and mood, and hyperarousal, as measured by changes in CAPS-5 subscale scores from Visit 3 (Baseline) to Visit 19 (18 weeks post Baseline)
- 3. Explore the effect of adverse childhood experiences (ACE) on the CAPS-5 Total Severity analyses
- 4. Explore changes in:
  - Dissociative symptoms associated with PTSD (DSP-I)
  - Depression (BDI-II)
  - Chronic pain (CPGS)
  - Quality of life (EQ-5D-5L)
  - Functioning in relation to self and others (IASC)
  - Psychosocial functioning (IPF)
  - Self-compassion (SCS)
  - Alexithymia (TAS-20)
  - Addictive behaviors including: alcohol use (AUDIT), drug use (DUDIT), and nicotine use (SRNU)
  - Eating habits (EAT-26)
  - Workplace productivity (HPQSF)
  - Healthcare utilization (UFEC)

5. Characterize the sample and effects of treatment on different outcomes

#### 4.0 Measures

## 4.1 Primary Measure

☐ Clinician Administered PTSD Scale for DSM-5 (CAPS-5)

## **4.2 Secondary Outcome Measure**

• Sheehan Disability Scale (SDS)

## 4.3 Safety Measures

| ] '] | l'rea | tment | t-emer | gent . | Ad | verse | event | ts |
|------|-------|-------|--------|--------|----|-------|-------|----|
|------|-------|-------|--------|--------|----|-------|-------|----|

☐ Concomitant medication use

☐ Vitals signs during MDMA sessions

☐ Columbia Suicide Severity Rating Scale (C-SSRS)

## **4.4 Exploratory Measures**

| Life | Events | Check | list | (LEC | C-5) | ) |
|------|--------|-------|------|------|------|---|
|------|--------|-------|------|------|------|---|

☐ Adverse Childhood Experience Questionnaire (ACE)

☐ Inventory of Psychosocial Functioning (IPF)

☐ The Dissociative Subtype of PTSD Interview (DSP-I)

☐ Beck Depression Inventory II (BDI-II)

☐ Chronic Pain Grade Scale (CPGS)

☐ Inventory of Altered Self Capacities (IASC)

☐ Toronto Alexithymia Scale (TAS-20)

☐ Self-Compassion Scale (SCS)

☐ EuroQol Five Dimensions – Five Levels Questionnaire (EQ-5D-5L)

☐ Eating Attitudes Test (EAT-26)

☐ Alcohol Use Disorders Identification Test (AUDIT)

☐ Drug Use Disorders Identification Test (DUDIT)

☐ Self-reported Nicotine Use (SRNU)

☐ Utilization of Facility-based and Emergent Care (UFEC)

☐ Health and Work Performance Absenteeism and Presenteeism Short Form (HPQSF)

## 5.0 Study Design

**Table 1: Dose Regimen of MDMA** 

| Tubic 1. Dos | Tuble 1. Dose Regimen of Wild Will | | |
|---|---|---|---|
| Experimental | <b>Initial Dose</b> | Supplemental Dose* | Min-Max Cumulative Dose |
| Session | | | |
| 1 | 100 mg | 50 mg | 100 mg to 150 mg |
| 2 | 100 or 125* mg | 50 or 62.5 mg | 100 mg to 187.5 mg |
| 3 | 100 or 125* mg | 50 or 62.5 mg | 100 mg to 187.5 mg |
| | | Total Cumulative Dose | 300 mg to 525 mg |

<sup>\*</sup> Unless contraindicated

**Table 2: Time and Events – Study Procedures** 

| | | | ing Period<br>weeks) | | Preparatory Period w/ Enrollment Confirmation (2-11 weeks) | | | |
|---|---|---|---|---|---|---|---|---|
| | | Screening | | Enrollment<br>V0 | Prepa | ratory | Baseline<br>CAPS-5 T1 | Baseline & Enrollment<br>Confirmation |
| Visit | Phone<br>Screening | Screening | IR Screening | | V1 | V2 | V3 | V4 |
| Visit Description | Phone<br>Calls | In-person<br>Visits & Labs | Telemedicine | Enrollment | Prep. 1 | Prep. 2 | Telemedicine | Prep. 3 & Enrollment<br>Confirmation |
| Visit Timing | Prior to Initial<br>Screening | Over 3 wks<br>(-2 weeks/+1<br>wks) | 2 days after<br>initial<br>eligibility met<br>(+7 days) | 2 days post IR<br>Screening<br>(+12 days) | Within 1 wk<br>of V0 (0 to<br>12 days) | Within 3 wks<br>of V1 | Post V2 &<br>Taper | Within 6 days of V3 |
| Initial Phone Screen | <b>√</b> | | | | | | | |
| Informed Consent | Send Copy | <b>√</b> | | | | | | |
| Follow-up Phone Screen | <b>√</b> | | | | | | | |
| Assess Eligibility | <b>√</b> | <b>√</b> | | ✓ | ✓ | ✓ | | ✓ |
| Medical/Psychiatric History | ✓ A | <b>√</b> | | | ✓ | ✓ | | ✓ |
| Past/Current Medication & Adherence | <b>√</b> | <b>√</b> | | | ✓ | ✓ | | ✓ |
| Weight, Resting Vitals | | <b>✓</b> | | | | | | |
| Physical Exam | | <b>√</b> | | | | | | |
| ECG & Rhythm Strip | | <b>√</b> | | | | | | |
| Clinical Lab Tests | | <b>√</b> | | | | | | |
| Drug Screen | | <b>√</b> | | | | | | <b>√</b> |
| Pregnancy Screen | | <b>√</b> | | | | | | <b>√</b> |
| Enter Participant in eCRF <sup>B</sup> | | <b>√</b> | | | | | | |
| Record | | | ✓ | | <b>√</b> | ✓ | <b>√</b> | <b>√</b> |
| Medication Taper | | | | ✓ | <b>√</b> | ✓ | | |
| Study Enrollment | | | | ✓ | | | | ✓ Confirmed |
| All AEs <sup>C</sup> | | | | ✓ | <b>√</b> | ✓ | | ✓ |
| 90-min Preparatory Session | | | | | <b>√</b> | <b>√</b> | | ✓ |
| Phone Call Follow-up D | _ | | | | | ✓ | | |

At Screening, collect data on previous hospitalizations and healthcare utilization. Request participants to obtain medical/psychiatric records to bring to the in-person screening.

B Participants will be entered into the eCRF after the IR visit is scheduled

C All Adverse Events (AEs) includes collecting Serious Adverse Events, AEs of Special Interest, AEs of Psychiatric Status, AEs requiring medical advice or attention, AEs that indicate withdrawal of a participant, and all other AEs

<sup>&</sup>lt;sup>D</sup> If needed, call participant to confirm medication tapering and stabilization is complete prior to Visit 3

| | | Treatment Period ~12 weeks (+/-3 weeks) | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Treatment 1 | | | | | | Treatmer | nt 2 | | | Treat | | Primary<br>Outcome | Study<br>Termi-<br>nation | |
| Visit | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | V18 | V19 | V20 |
| Visit Description | Exp. 1 | Int. 1.1 | Int.<br>1.2 | CAPS-5<br>T2: Tele-<br>medicine | Int. 1.3 | Exp. 2 | Int. 2.1 | Int.<br>2.2 | CAPS-5<br>T3: Tele-<br>medicine | Int. 2.3 | Exp. 3 | Int. 3.1 | Int. 3.2 | Int. 3.3 | CAPS-5<br>T4<br>Outcome:<br>Tele-<br>medicine <sup>H</sup> | Study<br>Termi-<br>nation |
| Visit Timing | Within<br>1 wk of<br>V3 | Morn-<br>ing<br>after<br>V5 | Within 2<br>wks<br>of V5 | Within 3<br>weeks<br>after V5 | 1-7<br>days<br>before<br>V10 | Within<br>4 wks<br>of V5<br>(+/-1<br>wk) | Morn-<br>ing<br>after<br>V10 | Within 2 wks of V10 | Within 3<br>weeks<br>after<br>V10 | 1-7 days<br>before<br>V15 | Within<br>4 wks<br>of V10<br>(+/-1<br>wk) | Morn-<br>ing<br>after<br>V15 | Within<br>2 wks<br>of V15 | Within<br>4 wks<br>of V15 | 8 wks<br>post V15<br>(+/-2 wk) | 2 days<br>post<br>V19 (-<br>1/+7<br>days) |
| Past/Current | | | | | | | | | | | | | | | | |
| Medication & | <b>√</b> | ✓ | <b>✓</b> | | ✓ | ✓ | ✓ | ✓ | | $\checkmark$ | <b>√</b> | ✓ | ✓ | ✓ | | ✓ |
| Adherence<br>Drug Screen | _ | | | | | _ | | | | | <b>✓</b> | | | | | |
| Pregnancy Screen | · / | | | | | · / | | | | | · / | | | | | |
| Record | · / | | _ | <b>√</b> | <b>√</b> | · / | | <b>√</b> | | <b>√</b> | · / | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | |
| All AEs C | · / | · · | · · | • | · / | · / | · / | · / | • | · / | · / | | · / | · / | • | <b>✓</b> |
| Container Assignment D | <b>✓</b> | | | | | <b>√</b> | | | | | <b>✓</b> | | | | | |
| Administer IP | <b>√</b> | | | | | <b>√</b> | | | | | <b>√</b> | | | | | |
| 8-hour Exp.<br>Session | ✓ | | | | | ✓ | | | | | ✓ | | | | | |
| BP, Pulse,<br>Temperature <sup>E</sup> | ✓ | | | | | ✓ | | | | | <b>√</b> | | | | | ✓ F |
| Overnight Stay I | <b>√</b> | | | | | ✓ | | | | | <b>✓</b> | | | | | |
| 90-min Integrative<br>Session | | ✓ | <b>✓</b> | | ✓ | | ✓ | ✓ | | ✓ | | ✓ | ✓ | ✓ | | |
| Phone Call<br>Follow-up <sup>G</sup> | | <b>✓</b> | | | | | <b>✓</b> | | | | | ✓ | | | | |
| Weight | | | | | | | | | | | | | | | | <b>✓</b> |

<sup>&</sup>lt;sup>C</sup> All Adverse Events (AEs) includes collecting Serious Adverse Events, AEs of Special Interest, AEs of Psychiatric Status, AEs requiring medical advice or attention, AEs that indicate withdrawal of a participant, and all other AEs

<sup>&</sup>lt;sup>D</sup> Obtain container assignment 24 to 48 hours prior to each Experimental Session

<sup>&</sup>lt;sup>E</sup> During Experimental Sessions, vitals are measured before Investigational Product administration, immediately before the supplemental dose is administered (or would be, if supplemental dose not given), and approximately 8 hours after initial dose, and as needed

F At Study Termination, only blood pressure needs to be measured

<sup>&</sup>lt;sup>G</sup> 4 days of phone call follow-up: Day 2 and 7 after the Experimental Session, with two additional calls in between

HAll visits must be scheduled to ensure that the Primary Outcome CAPS-5 T4 assessment is within the overall window provided: 18 weeks (+/-3 weeks) post V3

**Table 3: Time and Events – Study Measures** 

| | | Screening | | Baselin<br>Enrolln<br>Confirm | nent | | Treat | ment 1 | | Treatment 2 | | | | | reatment 3 | | Follow-up & Study<br>Termination | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit # | Site A | IR Screening | IR<br>V3 | V4 | V5 | V6&7 | IR<br>V8 | V9 | V10 | V11&12 | IR<br>V13 | V14 | V15 | V16&17 | V18 | IR<br>V19 | V20 |
| Visit Description | ~Time to<br>Complete<br>Measure<br>(minutes) | Site Visit | Tele-<br>medicine | Tele-<br>medicine | Site<br>Visit | Exp.<br>Session<br>1 | Int.<br>Sessions<br>1.1 &<br>1.2 | CAPS-5<br>T2: Tele-<br>medicine | | Exp.<br>Session 2 | Int.<br>Sessions<br>2.1 &<br>2.2 | CAPS-5<br>T3: Tele-<br>medicine | Int.<br>Session<br>2.3 | Exp.<br>Session 3 | Int.<br>Sessions<br>3.1 & 3.2 | Int.<br>Session<br>3.3 | CAPS-5<br>T4:<br>Outcome:<br>Tele-<br>medicine | Study<br>Termi-<br>nation |
| CAPS-5 | 90 (Baseline)<br>60 (all others) | | | <b>~</b> | | | | <b>\</b> | | | | <b>✓</b> | | | | | <b>√</b> | |
| SDS | 2 | | | <b>✓</b> | | | | <b>√</b> | | | | ✓ | | | | | ✓ | |
| DSP-I | 15 | | | ✓ | | | | ✓ | | | | ✓ | | | | | <b>√</b> | |
| C-SSRS B | 10 | <b>√</b> | <b>✓</b> | | <b>✓</b> | √c | ✓ | | ✓ | √c | ✓ | | ✓ | √c | <b>√</b> | ✓ | | <b>√</b> |
| MINI | 15 | | <b>✓</b> | | | | | | | | | | | | | | | |
| SCID-5-SPQ | 20 | <b>√</b> | | | | | | | | | | | | | | | | |
| SCID-5-PD | 60 | | ✓ | | | | | | | | | | | | | | | |
| LEC-5 | 5 | ✓ | | | | | | | <b>√</b> | | | | <b>✓</b> | | | ✓ | | <b>√</b> |
| PCL-5 | 8 | <b>√</b> | | | ✓ | | | | ✓ | | | | ✓ | | | | | <b>√</b> |
| DDIS D | 5 | | <b>√</b> | | | | | | | | | | | | | | | |
| ACE | 4 | | | | ✓ | | | | | | | | | | | | | |
| BDI-II | 10 (Baseline)<br>5 (all others) | | | | <b>√</b> | | | | | | | | | | | | | <b>√</b> |
| CPGS | 5 | | | | ✓ | | | | | | | | | | | | | <b>√</b> |
| EQ-5D-5L | 3 | | | | ✓ | | | | | | | | | | | | | <b>√</b> |
| IASC | 15 | | | | ✓ | | | | | | | | | | | | | ✓ |
| IPF | 10 | | | | ✓ | | | | | | | | | | | | | <b>√</b> |
| SCS | 6 | | | | <b>✓</b> | | | | | | | | | | | | | <b>√</b> |
| TAS-20 | 5 | | | | ✓ | | | | | | | | | | | | | ✓ |
| AUDIT | 3 | <b>✓</b> | | | | | | | | | | | | | | | | <b>√</b> |
| DUDIT | 3 | <b>✓</b> | | | | | | | | | | | | | | | | <b>√</b> |
| SRNU | 3 | | | | ✓ | | | | | | | | | | | | | <b>√</b> |
| EAT-26 | 6 | | | | ✓ | | | | | | | | | | | | | <b>√</b> |
| HPQSF | 5 | | | | ✓ | | | | | | | | | | | | | <b>√</b> |
| UFEC | 3 | | | | ✓ | | | | | | | | | | | | | |
| ~Total Time of Con<br>Measures (minutes | | 49 | 90 | 107 | 93 | 40 | 10 | 77 | 23 | 40 | 10 | 77 | 23 | 40 | 10 | 15 | 77 | 95 |

<sup>&</sup>lt;sup>A</sup> Ensure that LEC-5 and SCID-5-SPQ results are sent to the Independent Rater who will be conducting the SCID-5-PD

<sup>&</sup>lt;sup>1</sup>See Appendix A for exceptions to overnight stay directive

<sup>&</sup>lt;sup>B</sup> First C-SSRS is a Lifetime assessment, other assessments are Since Last Visit

<sup>&</sup>lt;sup>C</sup> Conducted pre- and post-Investigational Product administration, and at phone calls on Days 2 and 7 after Experimental Session

<sup>&</sup>lt;sup>D</sup> The relevant questions (117-130) from the DDIS will be asked by the Independent Rater during the SCID-5-PD assessment. The entire measure will never be administered.

## 6.0 Randomization and Blinding

MP17 is an open-label study with no randomization or blinding of treatment.

## 7.0 Sample Size and Power Considerations

MP17 is a one-arm interventional study. Thus, no power nor sample size calculations were required.

#### 8.0 Analyses

Every effort will be made to ensure complete, accurate and timely data collection and to avoid missing data, to ensure the completeness of the data which can impact the integrity and accuracy of the final study analysis. The statistical analyses will be reported using summary tables, figures, and data listings. All analyses and tabulations will be performed using SAS® Version 9.4 or higher, and S-PLUS. In general, nominal variables will be described in terms of frequencies and percentages. Ordinal and non-normal continuous variables will be described using sample median and range.

Approximately normal variables will be described using sample mean and standard deviations and analyzed by parametric statistical tests. Except for the primary effectiveness analysis, all statistical tests will be two-sided and a difference resulting in a p-value of less than or equal to 0.05 will be considered statistically significant. All p-values will be rounded to and displayed in four decimals. If a p-value less than 0.0001 occurs it will be shown in tables as <0.0001. Data not subject to analysis according to this plan will not appear in any tables or graphs, but will be included in the data listings. Selected results may be presented graphically using standard graphical software.

#### 8.1 Analysis Sets

- Safety: all participants who receive any IP
- All Enrolled: all participants who signed informed consent
- *Modified Intent-To-Treat (mITT):* all randomized participants who receive IP in at least one blinded Experimental Session (Visit 5) and have at least one follow-up CAPS-5 assessment post-treatment
- Per Protocol (PP): all randomized participants who meet eligibility criteria, who receive IP in three Experimental Sessions, and have three follow-up CAPS-5 assessments posttreatment
- Not Per Protocol (NPP): all participants who are included in the mITT set but not the PP set

#### 8.2 Missing Data Handling

All possible procedures within Good Clinical Practice (GCP) will be used to minimize Post-dosing Early Termination. Based on Phase 2 data it is expected that up to 5% of enrolled and

randomized participants will terminate early. Post-dosing Early Terminators will be compared to the Completers using baseline demographics and CAPS-5 Total Severity Score at baseline. Participants who are removed from the study after they are enrolled and receive IP but do not complete the study may fall into one of these categories: Post-Dosing Early Termination or Dropout. If the participant has received IP in at least one Experimental Session and completed one CAPS-5 assessment beyond Baseline, they will be considered evaluable. All participants who receive IP in at least one Experimental Session will be included in all safety analyses. Post-Dosing Early Termination are participants who discontinue study treatment but continue to participate in study evaluations and outcome assessments. Data collection by IRs will continue on the same schedule as planned through Study Termination visit procedures. Dropouts are defined as a participant who decides to withdraw consent. They will terminate without further follow-up. If the participant agrees, they will complete a final CAPS-5 assessment and Study Termination visit procedures. These participants are defined as dropouts who withdraw consent due to any reason after receiving at least one dose of IP and no longer participate in the study, i.e. no further contact with investigators or site staff. Data collected on study participants up to the time of withdrawal of consent will remain in the trial database in order to maintain scientific validity. Removal of data from the database would undermine the scientific and ethical integrity of the research. All observed CAPS-5 data up to the point of discontinuation of treatment will be included in the MMRM model of the *de jure* estimand from Post-dosing Early Terminators. Participants will not be replaced. All observed CAPS-5 data from Post-dosing Early Terminators and Dropouts collected prior to and after early termination will be included in the supportive effectiveness analysis of the de facto estimand.

## **8.2.1 Partial or Missing Dates**

The following conventions will be used to impute missing portions of dates for AEs and concomitant medications. Note that the imputed values outlined here may not always provide the most conservative date. In those circumstances, the imputed value may be replaced by a date that will lead to a more conservative analysis.

#### Start Dates:

- 1. If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- 2. If the month is unknown, then:
  - a. The month and day of the first dose date will be imputed if the year matches the first dose date year.
  - b. Otherwise, 'January' will be assigned.
- 3. If the day is unknown, then:
  - a. The day of the first dose date will be imputed if the month and year match the first dose date month and year.
  - b. Otherwise, the first day of the month will be assigned.

#### Stop Dates:

- 1. If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- 2. If the month is unknown, then 'December' will be assigned.
- 3. If the day is unknown, then the last day of the month will be assigned.

#### **8.3 Protocol Deviations**

A major deviation will be defined as participants enrolled and randomized but did not meet eligibility criteria during the course of the study, or any deviations that affect safety or overall data integrity, particularly if it relates to study endpoints. The number of participants in each protocol deviation category listed below will be summarized by analysis set and treatment group. Individual participants will appear in a listing.

Possible protocol deviations include the following categories:

- Participant entered study but did not meet criteria
- Participant developed withdrawal criteria but was not withdrawn
- Participant received excluded concomitant treatment
- Protocol procedure not performed per protocol
- Participant received incorrect treatment or incorrect dose
- Protocol procedure performed out of range
- Miscellaneous

#### 8.4 Baseline Values

Baseline values are from Baseline Visits for all measures, except C-SSRS, AUDIT, DUDIT, resting blood pressure (BP), Body Mass Index (BMI). For C-SSRS, the initial screening visit will be conducted with the 'Lifetime' version of the measure. The Independent Rater Screening assessment of 'Since Last Visit' suicidal ideation and behavior will be used as 'Baseline.' For the AUDIT and DUDIT measures and resting BP, BMI, results collected at Screening will be used as the Baseline value.

#### 8.5 Participant Disposition and Dosing Summary

The Safety Set will be included in the summary of participant disposition and accountability. The number and percent of participants who completed or discontinued the study will be displayed with reasons for early termination, where the percent is with respect to the total number of participants. The timepoint of doses and total MDMA (mg) administered will be summarized for the Safety Set.

#### 8.6 Demographics and Baseline Characteristics

Participant demographic data and Baseline characteristics will be summarized descriptively. The demographic data and baseline characteristics will be summarized for the Safety Set.

## 8.7 Effectiveness Analyses

For all primary, secondary, and exploratory endpoints descriptive statistics (n, mean, standard deviation, median, range, or counts and percentages where appropriate) will be provided. Longitudinal CAPS-5 Total Severity Score and SDS item scores will be plotted across visits to characterize the onset of treatment effect.

#### **8.7.1 Primary Effectiveness Analyses**

The *de jure* estimand of treatment effectiveness will be used to estimate the change in CAPS-5 score from baseline due to MDMA-assisted psychotherapy on PTSD symptom severity in the intended population of patients with PTSD from any cause. The primary estimator of effect will be the mean change in CAPS-5 Total Severity Scores from Baseline to 18 weeks after randomization (Visit 19). Least squares means from a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM) will be used to estimate the change in CAPS-5 from baseline to each visit. CAPS-5 data collected after treatment

discontinuation will not be included in the *de jure* estimand. Missing data will not be imputed.

## 8.7.2 Key Secondary Effectiveness Analyses

For the key secondary analysis of effectiveness, the de jure estimand will be used to estimate the estimate the change from baseline due to MDMA-assisted psychotherapy on PTSD on the SDS in the intended population of patients with PTSD from any cause. The SDS is a 3-item scale measuring the severity of disability in the domains of work, family life/home responsibilities and social/leisure activities. Each of these three domains is scored on a ten-point Likert scale, where a score of 0 is 'not at all impaired', 5 is 'moderately impaired' and 10 is 'very severely impaired'. For each study participant at each visit, the responses on the 3 items of the SDS will be summarized with a mean. In cases where the response on item 1 is not applicable, it will not be considered missing data. Thus, missing data assumptions and methodologies are not required when item 1 is not answered. Whereas when all 3 items have a response, the summary measure is the mean of the 3 item responses, in the cases where item 1 is not answered the summary measure will consist of the mean of items 2 and 3. It is expected that no more than 20% participants will have not have an applicable score for item 1, based on prior studies of paroxetine with PTSD. To limit missing data and ensure standardized administration, the SDS will be administered in a clinician-rated format during the same visits as the CAPS-5 by the centralized Independent Rater Pool.

The primary estimator of effectiveness will be the mean change in SDS Mean Scores from Baseline to 18 weeks after randomization (Visit 19). Least squares means from a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM) will be used to estimate the change from baseline to each visit. SDS data collected after treatment discontinuation will not be included in the *de jure* estimand. Missing data will not be imputed and will be considered missing at random.

#### 8.7.3 Exploratory Analyses

Post-hoc exploratory analyses not identified in this SAP may be performed to further examine the study data. These analyses will be clearly identified as such in the final clinical study report.

In exploratory analyses, additional baseline covariates (age, gender, ethnicity, index trauma, complexity and severity of trauma, medication tapering, diagnosis of comorbid depression, diagnosis of comorbid Axis 2 diagnosis, adverse childhood experiences) may be assessed for inclusion in the model at a p<0.05. One-group pretest-posttest Cohen's d effect size will be estimated.

#### 8.7.4 Responder Analyses

The CAPS-5 produces a Total Severity Score based on severity of PTSD symptom domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. A psychometric validation study found the following severity score ranges for the CAPS-5: Asymptomatic (0-10), Mild (11-22), Moderate (23-34), Severe (35-46), Extreme (47+). Based on these data, a 10-point reduction in CAPS-5 Total Severity Score is clinically meaningful. As an alternate definition of treatment response to assess clinical significance of study outcomes, the sponsor will conduct a responder analysis to support findings from the primary effectiveness analysis, and to explore how many single-dose treatments are needed to achieve response (See Figure 1).

Figure 1: CONSORT for PTSD Responder Analysis After Treatment



[1] Response at T2, T3, and T4 will be in comparison to Baseline at T1.

# 8.8 Safety Analyses

Safety assessment analyses for this study will include summaries of unsolicited adverse events, concomitant medications, suicidal ideation and behavior, and vital signs. Qualitative safety analyses will examine safety data with summary tables listing drug exposure, concomitant medications/therapies, unsolicited AEs, and percentages tabulated.

MP17 SAP

Version 2: 03 September 2019

## 8.8.1 Analysis of Exposure

The frequencies and percentages of participants with exposure will be summarized. Data will be tabulated for the Safety Set.

#### 8.8.2 Analysis of Adverse Events

The primary measure of safety will be the reporting of unsolicited AEs. All AEs collected from Enrollment to Termination will be categorized as follows:

- Pretreatment AEs are defined as AEs that occur during the Preparatory Period prior to the first dose in the first Experimental Session
- Treatment Emergent AEs are defined as AEs that occur during the Treatment Period from the first Experimental Session to the last Integrative Session
- AEs that occur on and two days after MDMA or placebo administration
- AESIs are defined as AEs specified in the protocol related to cardiac function and abuse liability
- Follow-up Period AEs are defined as AEs that occur during the Follow-up Period after the last Integrative Session through Termination
- AEs leading to discontinuation of IP
- AEs resulting in death or hospitalization.
- SAEs
- AEs continuing at Termination.

Verbatim terms on case report forms will be mapped to preferred terms (PT) and system organ class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA) Version 17.0. Frequency and incidence of AEs will be displayed by PT, sorted by SOC, and summarized by treatment group, analysis set, category (as defined above), severity, and seriousness. AEs will be analyzed and presented as follows:

- If a participant has more than one AE mapped to the same PT, that AE will be reported once using the highest severity
- Relationship will be determined based on relative incidence of TEAEs with at least two-fold difference between MDMA vs. placebo
- Compare relative incidence of AEs during Experimental Sessions such as clinical signs
  and symptoms, such as chest pain, shortness of breath, or neurological symptoms or
  any other signs or symptoms that may be indicative of a medical complication of the
  investigational product
- AEs that occur on day of Experimental Sessions and two days after IP administration will be presented separately.

#### 8.8.3 Concomitant Medications

A secondary measure of safety will be the reporting of concomitant medications. All concomitant medications collected from Screening to Study Termination will be categorized as follows:

- Pretreatment medications are defined as medications taken prior to and after signing informed consent and those taken during the Preparatory Period prior to the first Experimental Session. A stop date is expected prior to the first Experimental Session for any medications requiring a change in dose, a skipped dose, or tapering.
- Treatment Period concomitant medications are defined as those taken or continued during
  the Treatment Period from the first Experimental Session to the last Integrative Session.
  A stop date is expected prior to the each Experimental Session for any medications
  requiring a change in dose, a skipped dose, or tapering.
- Concomitant medications with a start date of the day of and two days after IP administration
- Follow-up Period concomitant medications are defined as those taken or continued during the Follow-up Period after the last Integrative Session through Termination
- Any concomitant medications that are tapered
- Any concomitant medications that are taken to treat an AE
- Any concomitant medications that are taken to treat an SAE
- Any excluded concomitant medications taken as a deviation from the protocol.

Concomitant medications on case report forms will be classified using the WHO Drug Dictionary Enhanced<sup>TM</sup> (WHO DDE). Frequency and incidence of concomitant medications will be displayed by generic name, sorted by class, and summarized by treatment group, analysis set, and category as defined above. Concomitant medications will be analyzed and presented as follows:

- Concomitant medications taken on the day of and two days after IP administration will be presented separately
- Any psychiatric concomitant medications by period.

#### 8.8.4 Analysis of Suicidal Ideation and Behavior

Suicidal ideation and behavior will be summarized according to suggestions made in the C-SSRS Scoring and Data Analysis Guide [1]. A positive response for suicidal ideation is counted when a participant answers "yes" to any one of the five suicidal ideation questions (Categories 1-5) on the C-SSRS (i.e., a score >0 for suicidal ideation). Serious suicidal ideation is a suicidal ideation score of 4 or 5. A positive response for suicidal behavior occurs when a participant answers "yes" to any one of the five suicidal behavior questions (Categories 6-10) on the C-SSRS (i.e., a score >0 for suicidal behavior). The number and percent of positive responses of Positive Ideation, Serious Ideation, and Positive Behavior will be tabulated by treatment group and time period (lifetime, screening, baseline, each Experimental Session (pre- and post-IP), Integrative Sessions, and endpoints). Frequency and incidence of positive or serious ideation and suicidal behavior will be presented using descriptive statistics in tabular format.

## 8.8.5 Summary of Vital Signs

Vital signs (heart rate, BP, and body temperature) for Experimental Sessions will be summarized using descriptive statistics in tabular format listing values at pre-IP, prior to the supplemental dose, and at the end of each Experimental Session. Change from Baseline in vital signs will be presented.

#### 9.0 Timing of Analyses

Preliminary analyses and listing reviews will be ongoing throughout the studies to inform therapist supervision and assumptions made for upcoming Phase 3 trials. For clinical study

reports and publications, only locked database files will be used. The primary effectiveness analysis will be conducted after all participants complete Visit 20 and the database is locked.

#### References

1. Nilsson, M.E., et al., *Columbia Suicide Severity Rating Scale Scoring and Data Analysis Guide*, in *CSSRS Scoring Version 2.0*. 2013:\_
<a href="http://www.cssrs.columbia.edu/documents/ScoringandDataAnalysisGuide\_Feb2013.pdf">http://www.cssrs.columbia.edu/documents/ScoringandDataAnalysisGuide\_Feb2013.pdf</a>.

p. 1-13.